CLINICAL TRIAL: NCT05084703
Title: Reproducibility of Functional Shoulder Tests for the Return to Sport of Patients Operated on Previous Shoulder Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A03013-52
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Latarjet; Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients operated for previous shoulder instability (Experimental): Different functionnal test to be done
  Interventions: Other: Functional tests
- Healthy volunteer (Active Comparator): Different functionnal test to be done
  Interventions: Other: Functional tests

INTERVENTIONS:
Other: Functional tests — * Symmetry indices between the two limbs obtained thanks to the scores of the functional tests : Y balance test
  * Muscle endurance index obtained from functional test scores : Closed Kinetic Chain Upper Extremitie Stability test

SUMMARY:
The aim of this study is to assess whether the indicators outcome of these tests discriminate between different populations. In particular to compare populations with shoulders without any history of injury with a population that had undergone a reduction in glenohumeral instability by the Latarjet technique.

DETAILED DESCRIPTION:
The different objectives of this study are :

* To assess the intra- and intersessional reproducibility of functional shoulder tests
* To evaluate the influence of an anterior front stop using the Latarjet method on the functional profile of the shoulder compared to a healthy population.

ELIGIBILITY:
Inclusion Criteria:

Patient group :

* Male patient
* Between 18 and 30 years-old
* Occurrence of the injury requiring surgery during a sports activity
* Reduction of shoulder instability by the Latarjet technique
* Surgery performed by surgeon from Santy orthopedic center (Lyon)
* Patient's inclusion by decision of the surgeon during the 4 months postoperatively visit

Healthy volunteer group :

* Male patient
* Between 18 and 30 years-old
* Patient regularly practicing sport activity.

Both groups :

* Patient having signed an informed consent
* Affiliated subject or beneficiary of a social security scheme

Exclusion Criteria:

Patient group :

* Contra indication from surgeon
* Having another pathology in the upper limbs
* Present a constitutional hyperlaxity
* Have stiffness or recurrence of dislocation of the shoulder post-surgery

Healthy volunteer group :

* Report a history of upper extremity pain / injury within the past 12 months
* Report a history of orthopedic surgery on the upper limbs

All participants :

* Protected subject : adult under guardianship, guardianship or other legal protection, deprived of liberty by judicial or administrative decision
* pregnant woman, breastfeeding, parturient

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2022-04-26 (Estimated)

PRIMARY OUTCOMES:
Symmetry indices between the two limbs obtained thanks to the scores of the functional tests | 1 hour
  using the Y balance test
Muscle endurance index obtained from functional test scores | 1 hour
  Using : Closed Kinetic Chain Upper Extremitie Stability test

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France